CLINICAL TRIAL: NCT05707377
Title: A Phase 2/3, Multicenter, Randomized, Active-Controlled, Open-label Study to Evaluate the Efficacy and Safety of Zanubrutinib in Patients With Primary Membranous Nephropathy
Brief Title: A Study to Examine the Efficacy and Safety of Zanubrutinib Given to Adults With Primary Membranous Nephropathy
Acronym: ALMOND
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-309; 2022-501147-32-00 (Registry Identifier: EU CTIS); CTR20230546 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Primary Membranous Nephropathy
Keywords: BGB-3111; Zanubrutinib; BTKi
MeSH Terms: interventions — zanubrutinib; Tacrolimus

STUDY DESIGN:
Intervention Model Description: In Part I, participants will be assigned to one treatment group. After enrollment in Part I is complete, enrollment in Part 2 will start. In Part 2, participants will be randomly assigned to 1 of 3 treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Zanubrutinib High Dose (Experimental): Participants will receive zanubrutinib twice daily.
  Interventions: Drug: Zanubrutinib
- Part 2: Zanubrutinib High Dose (Experimental): Participants will receive zanubrutinib twice daily.
  Interventions: Drug: Zanubrutinib
- Part 2: Zanubrutinib Low Dose (Experimental): Participants will receive zanubrutinib once daily.
  Interventions: Drug: Zanubrutinib
- Part 2: Tacrolimus (Active Comparator): Participants will receive tacrolimus capsules twice daily for 64 weeks.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib capsules administered orally.
  Other Names: BGB-3111; Brukinsa
  Arms: Part 1: Zanubrutinib High Dose; Part 2: Zanubrutinib High Dose; Part 2: Zanubrutinib Low Dose
Drug: Tacrolimus — Tacrolimus capsules administered orally.
  Arms: Part 2: Tacrolimus

SUMMARY:
The primary objectives of this study are: In Part 1 to evaluate the efficacy of zanubrutinib as measured by proteinuria reduction, and in Part 2 to evaluate the efficacy of zanubrutinib compared with tacrolimus as measured by complete remission rate, in participants with primary membranous nephropathy (PMN) who are on optimal supportive care.

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed PMN within 5 years before the initial screening (ie, the day the informed consent is signed)
* UPCR (based on 24-hour urine collection) > 3.5 at initial screening and at confirmation assessment
* Treatment with a maximally tolerated or allowed dose of an angiotensin-converting enzyme inhibitor (ACEI) or angiotensin II receptor blocker (ARB) for ≥ 24 weeks before randomization (12 weeks before initiation of study drug for Part 1) and with adequate blood pressure control (blood pressure < 130/80 mmHg, measured on ≥ 2 occasions [not on the same day] within 4 weeks before the assignment of study treatment)
* Anti-PLA2R antibody > 50 RU/mL at confirmation assessment (Part 1 only)

Exclusion Criteria:

* Participants with a secondary cause of membranous nephropathy
* Type 1 or 2 diabetes mellitus with hemoglobin A1c (HbA1c) ≥ 7% at screening
* Severe renal disease as determined by rapid decline in eGFR (defined as > 15 mL/min/1.73m^2 within 24 weeks prior to randomization, not otherwise explained)
* A known history of a primary immunodeficiency or an underlying condition such as human immunodeficiency virus (HIV) infection or splenectomy that predisposes the participant to infections
* Patients at risk for tuberculosis at screening
* Known infection with serologic status reflecting active or chronic hepatitis B virus infection, or presence of hepatitis C virus antibody
* Severe hepatic insufficiency (Child-Pugh C)
* Clinically significant cardio-cerebrovascular diseases

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change from Baseline in Urine Protein Creatinine Ratio (UPCR) | Baseline and Week 24
Part 2: Number of Participants Achieving Complete Remission | Week 104
  Complete remission is defined as:
  UPCR (based on 24-hour urine collection) ≤ 0.3, AND a stable estimated glomerular filtration rate (eGFR) (remains unchanged or decreases by < 15% compared with the baseline)

SECONDARY OUTCOMES:
Part 1: Number of participants with Treatment Failure | Week 24
Part 1: Number of Participants with Immunological Response | Week 24
  Immunological response is defined as anti- phospholipase A2 receptor (PLA2R) antibody level reduced from baseline to less than 14 relative units (RU)/ml.
Part 1: Number of Participants with Complete Remission | Week 24, Week 52, Week 76, and Week 104
  A complete remission is defined as:
  UPCR (based on 24-hour urine collection) ≤ 0.3, AND a stable eGFR (remains unchanged or decreases by < 15% compared with the baseline)
Part 1: Number of Participants with Overall Remission | Week 24, Week 52, Week 76, and Week 104
  Participants with overall remission are those achieving either complete remission or partial remission
Part 1: Number of Participants with Relapse | Week 104
  A relapse is defined as reappearance of UPCR (based on 24-hour urine collection) > 3.5 after complete or partial remission
Part 1: Number Of Participants with Treatment-Emergent Adverse Events (TEAEs) | From the first dose of study drug and up to 30 days after study drug discontinuation; up to approximately 68 weeks
Part 2: Number of Participants with Overall Remission | Week 24, Week 52, Week 76, and Week 104
  Participants with overall remission are those achieving either complete remission or partial remission
Part 2: Number of Participants with Complete Remission | Week 24, Week 52, and Week 76
  A complete remission is defined as:
  UPCR (based on 24-hour urine collection) ≤ 0.3, AND a stable eGFR (remains unchanged or decreases by < 15% compared with the baseline)
Part 2: Number of participants with Treatment Failure | Week 24, Week 52, Week 76, and Week 104
Part 2: Time to First Complete Remission | Up to approximately 104 weeks
  Time to First Complete Remission is the time from the date of randomization to the date of the first complete remission
Part 2: Time to First Overall Remission | Up to approximately 104 weeks
  Time to first overall remission is the time from the date of randomization to the date of the first overall remission
Part 2: Number of Participants with Relapse | Week 104
  A relapse is defined as reappearance of UPCR (based on 24-hour urine collection) > 3.5 after complete or partial remission
Part 2: Time to First Relapse | Up to approximately 104 weeks
  Time to first relapse is the time from the date of first complete or partial remission to the date of the first relapse
Part 2: Health Related quality of Life (HRQoL) Using the Kidney Disease and Quality of Life instrument™ - 36 items (KDQoL-36) | Up to approximately 104 weeks
Part 2: Health Related quality of Life (HRQoL) Using European Quality of Life 5-Dimensions 5-Levels Health Questionnaire (EQ-5D-5L) | Up to approximately 104 weeks
Number of Participants with ≥ 30% Estimated Glomerular Filtration Rate (eGFR) Reduction from Baseline | Baseline, Week 52, and Week 104
Part 2: Number of Participants with TEAEs | From the first dose of study drug and up to 30 days after study drug discontinuation; up to approximately 68 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (51):
- United States (6):
  - Amicis Research Center, Northridge, California
  - Stanford University, Palo Alto, California
  - Intermed Consultants, Minneapolis, Minnesota
  - Kidney Specialist of Southern Nevada (Ksosn), Las Vegas, Nevada
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Carolina Nephrology, Spartanburg, South Carolina
- Brazil (2):
  - Instituto Pro Renal Brasil, Curitiba
  - Hcfmusp Hospital Das Clinicas Da Faculdade de Medicina Da Universidade de Sao Paulo, São Paulo
- Ott Healthcare, Inc (Corporate Medical Centre), Scarborough Village, Ontario, Canada
- China (31):
  - Beijing An Zhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Guizhou Provincial Peoples Hospital, Guiyang, Guizhou
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Peoples Hospital, Taiyuan, Shanxi
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
- Czechia (2):
  - Fakultni Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- Istscientifico Di Pavia, Fondazione Smaugeri, Irccs, Clinica Del Lavoro E Della Riabilitazione, Pavia, Italy
- Medical Company Llc, Grozny, Chechenskaya Respublika, Russia
- Turkey (Türkiye) (2):
  - Erciyes University Medical Faculty, Erciyes
  - Kocaeli University Research and Application Hospital Department of Nephrology, Kocaeli
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - St Heliers Hospital, Carlshalton
  - Royal Derby Hospital, Derby
  - Aintree University Hospital, Liverpool
  - Manchester Royal Infirmary, Manchester

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397